CLINICAL TRIAL: NCT00107549
Title: A Phase I, Open-Label Study to Evaluate the Safety and Tolerability of Recombinant HIV-1 Vaccines in HIV-1 Infected Young Adults With Control of HIV-1 Replication and on Stable Highly Active Antiretroviral Therapy (HAART)
Brief Title: Safety of Recombinant HIV Vaccines in HIV Infected Young Adults on Stable Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P1059; 10051 (Registry Identifier: DAIDS ES Registry Number); PACTG P1059
Record Dates: First submitted 2005-04-05; First posted 2005-04-06 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Treatment Experienced; HIV Therapeutic Vaccine
MeSH Terms: conditions — HIV Infections

ARMS (1):
- 1 (Experimental): All participants in this study will receive two injections of the rMVA-HIV vaccine and the rFPV-HIV vaccine
  Interventions: Biological: rMVA-HIV (env/gag [TBC-M358] + tat/rev/nef-RT [TBC-M335)]); Biological: rFPV-HIV (env/gag [TBC-F357] + tat/rev/nef-RT [TBC-F349])

INTERVENTIONS:
Biological: rMVA-HIV (env/gag [TBC-M358] + tat/rev/nef-RT [TBC-M335)]) — Recombinant experimental therapeutic vaccine using the modified vaccinia Ankara vector given at study entry and Week 4
Biological: rFPV-HIV (env/gag [TBC-F357] + tat/rev/nef-RT [TBC-F349]) — Recombinant experimental therapeutic vaccine using fowlpox vector given at Weeks 8 and 24

SUMMARY:
The purpose of this study is to determine the safety of two recombinant HIV vaccines in HIV infected young adults on stable anti-HIV therapy.

DETAILED DESCRIPTION:
By helping to control viral replication, HAART has dramatically improved the prognosis for HIV infected individuals. However, because of extensive side effects, some of which may be acute and life-threatening, many patients find it difficult to tolerate a HAART regimen. HAART-associated long-term morbidity or mortality contribute to this difficulty. Administering an HIV therapeutic vaccine might allow HIV infected individuals to delay or interrupt treatment, avoiding the side effects associated with antiretroviral exposure. This study will evaluate the safety of two injections of two recombinant therapeutic vaccines in HIV infected young adults who are currently on stable HAART.

This study will last 72 weeks. All participants will receive two rMVA vaccines (env/gag and tat/rev/nef-RT) at study entry and at Week 4 and two rFPV vaccines (env/gag and tat/rev/nef-RT) at Weeks 8 and 24. Safety will be assessed immediately after each immunization and at 1 hour and 48 hours postimmunization. There will be 16 study visits over 72 weeks. A physical exam, blood collection, and administration of an adherence module will occur at most visits. An electrocardiogram (ECG) will occur at study entry and Weeks 2 and 10. Urine collection will occur at study entry and Weeks 4, 8, and 24.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected
* CD4 count of 350 cells/mm3 or greater
* If hepatitis B or C infected, infection must be chronic and stable
* Normal electrocardiogram (ECG)
* On stable HAART consisting of at least 3 different antiretrovirals from 2 different classes AND with a viral load of less than 100 copies/ml for at least 6 months prior to study entry
* Willing to use acceptable forms of contraception. Females enrolled in the study must use contraception for at least 21 days prior to first vaccination until the last study visit. Males enrolled in the study must use a condom from the first vaccination until one month after the last vaccination.
* Willing to follow all study requirements
* Available for follow-up for the duration of the study

Exclusion Criteria:

* History of allergic reaction to eggs or egg products
* Known hypersensitivity to vaccine components
* Chemotherapy for active cancer in the 12 months prior to study entry
* Prior vaccination with any HIV-1 vaccine
* Prior vaccination against smallpox
* Prior vaccinia immunization
* Any immunization within 1 month of study screening
* History of or known active heart disease including myocardial infarction, angina pectoris, congestive heart failure, cardiomyopathy, pericarditis, stroke or transient ischemic attack, chest pain or shortness of breath with activity such as walking upstairs, mitral valve prolapse, or other heart conditions under a doctor's care
* Immunomodulatory agents, gamma globulin, or investigational agents within 6 months of study entry
* Systemic steroids, including nonprescription street steroids, within 6 months of study entry
* Documented or suspected serious bacterial infection, metabolic illness, cancer, or immediate life-threatening condition
* Any clinically significant diseases other than HIV infection or clinically significant findings during study screening that, in the investigator's opinion, may interfere with the study
* Current alcohol or drug abuse that, in the investigator's opinion, may interfere with the study
* Pregnancy or breastfeeding

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Development of any adverse events of Grade 3 or higher | Throughout study
Development of adverse events of Grade 3 or higher attributed to the study vaccines | Throughout study
Viral breakthrough to greater than 1,000 copies/ml | During the first 24 weeks of study

CONTACTS AND LOCATIONS:
Overall Officials: Coleen K. Cunningham, MD, Study Chair — Pediatric Infectious Diseases, Duke University
Locations (9):
- United States (8):
  - Children's Hospital Los Angeles NICHD CRS, Los Angeles, California
  - Usc La Nichd Crs, Los Angeles, California
  - Univ. of Colorado Denver NICHD CRS, Aurora, Colorado
  - Chicago Children's CRS, Chicago, Illinois
  - Univ. of Maryland Baltimore NICHD CRS, Baltimore, Maryland
  - Columbia IMPAACT CRS, New York, New York
  - DUMC Ped. CRS, Durham, North Carolina
  - St. Jude/UTHSC CRS, Memphis, Tennessee
- Univ. of Puerto Rico Ped. HIV/AIDS Research Program CRS, San Juan, Puerto Rico

REFERENCES:
- [Background] Caputo A, Gavioli R, Ensoli B. Recent advances in the development of HIV-1 Tat-based vaccines. Curr HIV Res. 2004 Oct;2(4):357-76. doi: 10.2174/1570162043350986. PMID 15544457
- [Background] Cosma A, Nagaraj R, Buhler S, Hinkula J, Busch DH, Sutter G, Goebel FD, Erfle V. Therapeutic vaccination with MVA-HIV-1 nef elicits Nef-specific T-helper cell responses in chronically HIV-1 infected individuals. Vaccine. 2003 Dec 8;22(1):21-9. doi: 10.1016/s0264-410x(03)00538-3. PMID 14604567
- [Background] Kent SJ, Zhao A, Best SJ, Chandler JD, Boyle DB, Ramshaw IA. Enhanced T-cell immunogenicity and protective efficacy of a human immunodeficiency virus type 1 vaccine regimen consisting of consecutive priming with DNA and boosting with recombinant fowlpox virus. J Virol. 1998 Dec;72(12):10180-8. doi: 10.1128/JVI.72.12.10180-10188.1998. PMID 9811759
- [Background] Mwau M, Cebere I, Sutton J, Chikoti P, Winstone N, Wee EG, Beattie T, Chen YH, Dorrell L, McShane H, Schmidt C, Brooks M, Patel S, Roberts J, Conlon C, Rowland-Jones SL, Bwayo JJ, McMichael AJ, Hanke T. A human immunodeficiency virus 1 (HIV-1) clade A vaccine in clinical trials: stimulation of HIV-specific T-cell responses by DNA and recombinant modified vaccinia virus Ankara (MVA) vaccines in humans. J Gen Virol. 2004 Apr;85(Pt 4):911-919. doi: 10.1099/vir.0.19701-0. PMID 15039533
- [Background] Pancharoen C, Ananworanich J, Thisyakorn U. Immunization for persons infected with human immunodeficiency virus. Curr HIV Res. 2004 Oct;2(4):293-9. doi: 10.2174/1570162043351084. PMID 15544450
- [Derived] Shiu C, Cunningham CK, Greenough T, Muresan P, Sanchez-Merino V, Carey V, Jackson JB, Ziemniak C, Fox L, Belzer M, Ray SC, Luzuriaga K, Persaud D; Pediatric AIDS Clinical Trials Group P1059 Team. Identification of ongoing human immunodeficiency virus type 1 (HIV-1) replication in residual viremia during recombinant HIV-1 poxvirus immunizations in patients with clinically undetectable viral loads on durable suppressive highly active antiretroviral therapy. J Virol. 2009 Oct;83(19):9731-42. doi: 10.1128/JVI.00570-09. Epub 2009 Jul 15. PMID 19605490